CLINICAL TRIAL: NCT05494957
Title: Clinical Study of New Intensive Treatment Regimen for Severe Nontuberculous Mycobacterial Pulmonary Disease
Acronym: NTM-PD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Shanghai Public Health Clinical Center (Other Government); No.85 Hospital, Changning, Shanghai, China (Other); Anhui Chest Hospital (Other); Shanghai Pudong New Area Pulmonary Hospital, China (Unknown); Huashan Hospital (Other); Zhengzhou Sixth People's Hospital, China (Unknown)
Responsible Party: Principal Investigator, Wei Sha MD & PhD, Director, Head of Tuberculosis Department,Shanghai Pulmonary Hospital, Principal Investigator, Clinical Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Q20-293
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Nontuberculous Mycobacterial Lung Disease
Keywords: Nontuberculous Mycobacterial Lung Disease; bedaquiline; Clofazimine

STUDY DESIGN:
Intervention Model Description: Treatment regimens containing bedaquiline, linezolid, clofazimine, and other drugs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New treatment regimen including bedaquiline (Experimental): Treatment regimens that include bedaquiline, linezolid, clofazimine, and other optional drugs.
  Interventions: Drug: New regimen(BdqCfzLzd+XY)

INTERVENTIONS:
Drug: New regimen(BdqCfzLzd+XY) — The basic regimen consists of bedaquiline, clofazimine, linezolid, and 2-3 drugs such as amikacin and tigecycline are selected according to the drug use history and in vitro culture drug sensitivity results to form the regimen, and the treatment period is usually more than 12 months, and the doses of various drugs are used for the regular drug use.
  Other Names: New regimen for NTM-PD(BdqCfzLzd+XY)

SUMMARY:
Investigators have selected a number of new drugs, including bedaquiline, to form a regimen to conduct clinical studies for the treatment of severe NTM lung disease.

DETAILED DESCRIPTION:
Currently, the annual prevalence of nontuberculous mycobacterial lung disease is increasing year by year. the clinical presentation of NTM is similar to that of tuberculosis, but most NTM is severely resistant to antibiotics, making it difficult to treat, and it responds poorly to classical antituberculous mycobacterial drugs. the overall response rate for the treatment of NTM lung disease is approximately 50% according to current domestic and international treatment guidelines. In severe NTM lung disease, after more than one anti-mycobacterial treatment, the resistance rate is even higher, the disease is more severe, and treatment is even more difficult. Current clinical treatment regimens are mainly long courses and combinations of drugs, however, the results are often unsatisfactory with an overall cure rate of only 30%. Therefore, we need to continue to explore new effective drugs for NTM lung disease and explore new and more effective drug regimens.

Several drugs have shown promising effects in basic research and clinical applications for NTM. For example, clofazimine has shown good efficacy in the treatment of nontuberculous mycobacterial lung disease. In addition, some new antibiotics or anti-tuberculosis drugs have attracted attention for showing good anti-NTM effects in in vitro experiments, such as tigecycline, linezolid, and bedaquiline. Based on the clinical experience of the investigators and related basic research, we conducted a clinical study of new regimens for intensive treatment of severe non-tuberculous mycobacterial lung disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-tuberculous mycobacterial lung disease who meet the diagnostic criteria of the American Thoracic Society and British Thoracic Society guidelines or the Chinese Expert Consensus on the Diagnosis and Treatment of Non-tuberculous Mycobacteriosis (2020) and whose strain is identified as Mycobacterium intracellulare/abscessus
2. Proposed anti-NTM therapy based on current disease.
3. Patients aged 18 to 65 years.
4. able to understand and have signed an informed consent form.
5. culture drug sensitivity results showing resistance to clarithromycin; or previous anti-NTM therapy has been ineffective.
6. Patients with severe NTM lung disease, with chest CT showing greater than 50% of the extent of infection lesions in both lungs; or with short-term progressive worsening of the disease.

Exclusion Criteria:

1. History of allergy to any drug in the protocol
2. Combined hepatic, renal, metabolic, autoimmune diseases, endocrine, hematological, neurological diseases, psychiatric disorders, malignancies, long-term immunosuppressive drugs or HIV/AIDS patients
3. QTc interval >470 ms in women and >450 ms in men
4. Severe pulmonary hypoplasia (FEV <30%)
5. Those with co-infection with other Mycobacterium species
6. Pregnant or breastfeeding females.
7. Those who are also participating in other clinical studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2022-08-05 (Estimated); Primary Completion 2024-08-05 (Estimated); Study Completion 2025-08-05 (Estimated)

PRIMARY OUTCOMES:
Treatment Outcome | Treatment period, approximately 12 months.
  Evaluation of treatment outcome at completion of treatment: can be classified as bacteriologically negative; bacteriologically cured; clinically cured; cured; treatment failure; bacteriological relapse; death.

SECONDARY OUTCOMES:
Improvement rate of imaging | Treatment period, approximately 12 months.
  Changes in imaging aspects of completed treatment compared to baseline can be classified as: absorption, significant absorption, no change, deterioration

OTHER OUTCOMES:
Improvement in lung function | Treatment period, approximately 12 months.
  Improvement of lung function FEV1 after treatment compared to baseline.
Adverse Events | Treatment period, approximately 12 months.
  Adverse Events that occurred during the study: Grade 3 or higher adverse reactions during treatment, or significant abnormalities in vital signs.
Mycobacterial culture negative conversion rate | Treatment period, approximately 12 months.
  Mycobacterial culture negative conversion rate at the end of the treatment course compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No